CLINICAL TRIAL: NCT00088569
Title: Measuring the Brain Effects of DC Polarization With O-15 PET
Brief Title: Effect of Direct Current Polarization on Brain Function
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040220; 04-N-0220
Record Dates: First submitted 2004-07-29; First posted 2004-07-30 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-06

CONDITIONS: Healthy
Keywords: Frontal Lobe; Working Memory; Treatment; Transcranial; Electrical; Healthy Volunteer; HV

INTERVENTIONS:
Drug: 0-15 Water

SUMMARY:
This study will test a new electrical technique called direct current (DC) polarization that is able to change brain activity in subtle ways for a short time. A recent study showed that, depending on its direction, the current could make people perform a little better or perhaps slightly worse on a test of the function of the brain's frontal lobe. This study will use positron emission tomography (PET) scanning to examine how DC polarization affects brain activity.

Healthy volunteers between 20 and 70 years of age who are right handed and who are not taking any medications that affect the brain may be eligible for this study. Candidates are screened with a brief medical history and neurological evaluation.

Participants have a PET scan on three different days at least 3 days apart. Each scanning session takes 2-1/2 to 3 hours. For the scan, radioactive water is injected into the body through a vein. Subjects lie on a bed that slides in and out of the doughnut-shaped scanner, with their head held from the back by a padded holder and in front by a custom-molded plastic mask with holes for the eyes, nose, and mouth. DC electrodes made of wet sponges are placed on the right side of the head and over the left eye and are held in place with elastic bandages.

Three kinds of DC polarization are tested. In two tests the current is the same, but in opposite directions. The third is a sham (placebo) condition with no current delivered. Each of the three scans is separated by at least 3 days. On each day, a series of scans is done in a single session. Before each injection of tracer, the DC current is turned on. This may cause a tingling or slight burning on the skin under the electrodes, which disappears when the current is turned off. In each session, the subject receives 16 injections of tracer about 8 minutes apart, with DC polarization turned on for 4 out of the 8 minutes.

During most of the 8-minute periods, subjects are shown a pattern of dots about every 2 seconds. Sometimes the subject just looks at the patterns, and sometimes subjects are asked to push a button corresponding to the pattern they saw just before the current one. Sometimes they will be asked to push a button corresponding to the pattern that came before that one and so on, up to three patterns before the current one. The task lasts for about 2 minutes each time, with time to relax in between.

DETAILED DESCRIPTION:
Objective: The passage of weak DC currents across the head (DC polarization) is a safe and painless means of altering the activity of cortical neurons and their response to exogenous stimulation. This has been demonstrated in the human motor cortex where local anodal polarization increases, and cathodal decreases, the motor evoked potential from TMS. Recent experiments from our lab suggest that polarization may have analogous effects on the prefrontal cortex, where anodal current enhances functions including verbal fluency and psychomotor speed and cathodal current produces slight performance decrements. We are interested in the potential of DC current to enhance function in patients with frontal lobe disorders and to reduce frontal overactivation in conditions such as drug craving. Treatments that alter frontal activity may also have mood altering properties. In order to establish the principle that DC polarization is able to alter frontal lobe activity we propose to combine DC polarization with a variably loaded frontal activation task and measure regional cerebral blood flow (rCBF with H(2)(15)O positron emission tomography (PET) scanning.

Study population: Twenty healthy individuals will be studied.

Design: On three different days, participants will receive right dorsolateral prefrontal anodal, cathodal, or sham treatment. On each day, rCBF will be measured during rest without and then with treatment. Then subjects will perform the N-back task (a test of working memory) during treatment with the working memory load (N) varied between 0 and 3 items from scan to scan.

Outcome measures: Resting rCBF and the relationship between cognitive load and rCBF at the treatment site will be compared between treatments in order to look for effects on task-related activation and performance.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants will be right-handed volunteers, aged 20 to 70, without history of any disorder of the central nervous system.

EXCLUSION CRITERIA:

Current serious medical or psychiatric condition of any kind.

History of any significant trauma or medical condition affecting the brain or skull.

History of epileptic seizure.

Current use of neuroactive medications, medications affecting the cerebral circulation, or recreational drugs.

Presence of metal in the head (other than dental hardware) or body, such as pacemakers, aneurysm clips, metallic prostheses (including heart valves or cochlear implants), patches with metallic foil backing, such as nicotine patches, permanent eyeliner or shrapnel fragments.

History of welding or metal work.

Broken skin in the area of the stimulating electrodes.

Pregnancy/breastfeeding.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Antal A, Kincses TZ, Nitsche MA, Paulus W. Modulation of moving phosphene thresholds by transcranial direct current stimulation of V1 in human. Neuropsychologia. 2003;41(13):1802-7. doi: 10.1016/s0028-3932(03)00181-7. PMID 14527543
- [Background] Antal A, Kincses TZ, Nitsche MA, Paulus W. Manipulation of phosphene thresholds by transcranial direct current stimulation in man. Exp Brain Res. 2003 Jun;150(3):375-8. doi: 10.1007/s00221-003-1459-8. Epub 2003 Apr 16. PMID 12698316
- [Background] Antal A, Kincses TZ, Nitsche MA, Bartfai O, Paulus W. Excitability changes induced in the human primary visual cortex by transcranial direct current stimulation: direct electrophysiological evidence. Invest Ophthalmol Vis Sci. 2004 Feb;45(2):702-7. doi: 10.1167/iovs.03-0688. PMID 14744917